CLINICAL TRIAL: NCT06862726
Title: Study of the Inter- and Intra-individual Variability of Anti-Xa Activity of Apixaban Versus Rivaroxaban Versus Control Arm During Non-valvular Atrial Fibrillation: Evaluation of Stability and Clinical Impact
Brief Title: Apixaban Versus Rivaroxaban in Non Valvular Atrial Fibrillation
Acronym: APIXA-Xa
Status: Enrolling by invitation | Phase: Phase 4 | Type: Interventional
Sponsor: Les Laboratoires des Médicaments Stériles (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Apixa Xa
Record Dates: First submitted 2024-11-25; First posted 2025-03-06 (Actual); Last update posted 2025-03-06 (Actual); Status verified 2025-02

CONDITIONS: Non Valvular Atrial Fibrillation
Keywords: non valvular atrial fibrillation; Direct oral anticoagulant; thromboembolic events; hemorrhage; anti-FXa activity; variability
MeSH Terms: conditions — Thromboembolism; Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- VKA (Active Comparator): This arm contain 40 patients on anti-vitamin K. Their prothromin level and INR will be measured
  Interventions: Drug: Dosage of PT-INR
- Apixaban (Active Comparator): This arm contain 40 patients. Anti Xa activity and Time in the range will be monitored
  Interventions: Drug: Anti Xa dosage
- Rivaroxaban (Active Comparator): This arm contain 40 patients. Anti Xa activity and Time in the range will be monitored
  Interventions: Drug: Anti Xa dosage

INTERVENTIONS:
Drug: Anti Xa dosage — VKA: quadriseparable tablet Apixaban: 5 mg twice daily or 2.5 twice daily Rivaroxaban: 20 mg once a day or 15 mg once a day
  Arms: Apixaban; Rivaroxaban
Drug: Dosage of PT-INR — This arm contain 40 pateints treated by VKA,. PT-INR dosage will be performed.
  Arms: VKA

SUMMARY:
The investigators will first measure the maximum concentration (after 2 hours of intake) and the residual concentration (just before the next intake) after at least 15 consecutive days of treatment.

In order to be able to study the stability of the anti-Xa activity of Apixaban vs Rivaroxaban, as well as their impact on the risk of thromboembolic events or hemorrhagic events, clinical follow-up and a determination of maximum and residual activity are necessary, ideally at 3 to 6 months (compared to studies carried out in the literature).

This evaluation would be made according to a multivariate analysis taking into consideration the other clinical-biological data relating to the patient, namely renal function, liver function, CHA2DS2-VASc score, HAS-BLEED score, treatment compliance, etc.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is the most common heart rhythm disorder with an estimated global prevalence of between 1 and 2%. It is a serious pathology that considerably increases morbidity and mortality. Thromboembolic events are a major complication .

Thus, effective anticoagulation is one of the major pillars of the management of atrial fibrillation. This anticoagulation was for a long time based on vitamin K antagonists (VKAs) which have proven their effectiveness in significantly reducing the risk of thromboembolic complications. However, VKAs have several drawbacks, mainly related to their narrow therapeutic range, their high inter-individual variability and their multiple drug interactions. As a result, the use of VKAs is restrictive because of the need for a delicate, regular and individual adjustment of the effective dose based on the result of the INR (need for regular and close biological monitoring) .

Since 2007, a new class of oral anticoagulant encompassing direct oral anticoagulants has emerged and is increasingly beginning to take the place of VKAs in several pathologies, including AF. Indeed, DOACs are currently the first-line treatment during AF thanks to the results of randomized controlled clinical trials that have proven an efficacy at least equivalent to VKA without increasing the risk of serious bleeding. In addition, DOACs are simpler to use compared to VKAs because of their predictable pharmacodynamics and pharmacokinetics, which make it possible to use a fixed dose and dispense with biological monitoring of their plasma levels in the majority of cases.

However, it seems that there is a significant inter- and intra-individual variability related to the use of DOACs. In addition, the theory of a single dose and the non-need for monitoring is beginning to be debated. Indeed, the indications requiring an AOD assay seem to be broadening. Recently, studies have been identified in the literature that are interested in assessing the impact of the maximum and residual activity of DOAC on its efficacy and safety. Despite significant results, especially in relation to the fluctuation of residual activity, there are so far no strong conclusions of a high level of evidence that can rule on the usefulness of adjusting the dose according to the dosage of activity.

ELIGIBILITY:
Inclusion Criteria:

* Male or female ≥ 18 years of age
* Patients diagnosed with AF;
* Written informed consent obtained prior to participation in the study.

Exclusion Criteria:

* Patients with at least one of the following criteria will not be included in the trial:
* History of hypersensitivity to study drugs or drugs with a similar chemical structure.
* Patients receiving combination therapy of P-glycoprotein inhibitors or inducers such as itraconazole, ketoconazole, voriconazole, posaconazole, ritonavir, rifampicin, phenytoin, phenobarbital, and carbamazepine, within 14 days prior to taking apixaban
* Pregnant women
* Breastfeeding
* Patients Enrolled in Other Clinical Studies
* Patients who refuse to sign consent.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare the variability of anti-FXa activity of apixaban versus rivaroxaban | 6 months
  The patient will attend an initial appointment between 2 and 4 weeks to undergo sampling and receive their samples, followed by further appointments at 3 and 6 months. During these visits, samples will be collected to measure the anti-Xa activity of rivaroxaban and apixaban.
  Each sampling will occur in two steps: the first sample will be taken before the morning dose to measure anti-Xa activity at the trough (or nadir), and the second sample will be collected 2 hours later to determine the peak (or maximum value reached). The results will be expressed in nanograms per milliliter (ng/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Charles Nicolle hospital, Tunis, Tunisia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mavri A, Vene N, Bozic-Mijovski M, Miklic M, Soderblom L, Pohanka A, Malmstrom RE, Antovic J. Apixaban concentration variability and relation to clinical outcomes in real-life patients with atrial fibrillation. Sci Rep. 2021 Jul 6;11(1):13908. doi: 10.1038/s41598-021-93372-9. PMID 34230559
- [Result] Katritsis DG, Gersh BJ, Camm AJ. Anticoagulation in Atrial Fibrillation - Current Concepts. Arrhythm Electrophysiol Rev. 2015 Aug;4(2):100-7. doi: 10.15420/aer.2015.04.02.100. PMID 26835109